CLINICAL TRIAL: NCT04198714
Title: The Effect of Pudendal Nerve Block Analgesia on Postoperative Pain Control in Patients Undergoing Vaginal Surgery: A Randomized Double-blind Placebo-controlled Trial
Brief Title: Pudendal Nerve Block in Vaginal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB18-00759
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Nerve Block; Pain, Postoperative; Pelvic Floor Disorders; Pelvic Organ Prolapse; Pudendal Neuralgia; Surgery
MeSH Terms: conditions — Pain, Postoperative; Pelvic Floor Disorders; Pelvic Organ Prolapse; Pudendal Neuralgia

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block (Experimental): 9cc of 0.25% Marcaine + 1cc of 40mg/mL triamcinolone. 5cc will be injected transvaginally in the area of the pudendal nerve on each side.
  Interventions: Procedure: Pudendal block
- Placebo injection (Placebo Comparator): 10cc normal saline. 5cc will be injected transvaginally in the area of the pudendal nerve on each side.
  Interventions: Procedure: Pudendal block

INTERVENTIONS:
Procedure: Pudendal block — Administration of a pudendal block at the conclusion of vaginal surgery.

SUMMARY:
The objective of this this randomized controlled study is to determine whether a pudendal nerve block at the time of vaginal surgery is associated with improved postoperative pain control and decrease opioid consumption compared to a sham pudendal nerve block in patients undergoing vaginal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consenting, English speaking women between ages 18 and 80 who will undergo vaginal surgery
* Ability to read VAS Scores
* Specific vaginal procedures include, but are not limited to:

Perineoplasty Complete vaginectomy Le Forte colpocleisis Anterior repair, posterior repair, and/or enterocele repair Transvaginal mesh use Transvaginal mesh excision Sacrospinous ligament fixation Uterosacral ligament suspension Vaginal paravaginal defect repair Midurethral sling placement Sphincteroplasty Vaginal hysterectomy, with or without removal of tube(s) and/or ovary(s), with or without repair of enterocele

Exclusion Criteria:

* History of chronic pelvic pain
* Currently taking sedatives
* Liver disease
* Renal disease
* Women who did not consent for the study.
* Intraoperative concern for increased blood loss
* Unable to speak English
* Unable to understand VAS Scores
* Undergoing concomitant abdominal or laparoscopic procedures
* Allergy to bupivacaine or triamcinolone
* Planned abdominal or laparoscopic procedures.
* Patients who are ineligible for non-narcotic pain medications, such as an allergy to acetaminophen or NSAIDs

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Le Neveu M, Sears S, Rhodes S, Slopnick E, Petrikovets A, Mangel J, Sheyn D. The Impact of Pudendal Nerve Injection in Vaginal Surgery: A Secondary Analysis. Urogynecology (Phila). 2025 Sep 1;31(9):857-864. doi: 10.1097/SPV.0000000000001565. PMID 39733282
- [Derived] Slopnick EA, Sears SB, Chapman GC, Sheyn DD, Abrams MK, Roberts KM, Pollard R, Mangel J. Pudendal Nerve Block Analgesia at the Time of Vaginal Surgery: A Randomized, Double-Blinded, Sham-Controlled Trial. Urogynecology (Phila). 2023 Oct 1;29(10):827-835. doi: 10.1097/SPV.0000000000001351. Epub 2023 Apr 4. PMID 37093572

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pudendal Block | Placebo Injection
Started | 36 | 36
Completed | 36 | 35
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pudendal Block: Medication arm, received 9cc 0.5% bupivacaine + 1cc 40mg/cc triamcinolone 5 cc injected on each side
- Placebo Injection: Placebo arm, received 10cc normal saline 5cc injected on each side
- Total: Total of all reporting groups
Arm/Group | Pudendal Block | Placebo Injection | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.69 (10.41) | 58.54 (13.18) | 59.89 (11.943)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian | 1 | 0 | 1
  Race/Ethnicity: Black | 5 | 8 | 13
  Race/Ethnicity: Hispanic | 2 | 1 | 3
  Race/Ethnicity: White | 28 | 24 | 52
  Race/Ethnicity: Note specified | 0 | 2 | 2
Obesity [Count of Participants; unit: Participants] | 12 | 15 | 27
Tobacco use [Count of Participants; unit: Participants] | 3 | 4 | 7
Chronic pain [Count of Participants; unit: Participants] | 6 | 7 | 13
Preoperative diagnosis [Count of Participants; unit: Participants]
  Pelvic organ prolapse | 33 | 35 | 68
  Urinary incontinence | 18 | 14 | 32
  Vaginal mesh exposure | 1 | 0 | 1
  Uterine fibroids | 2 | 0 | 2
Surgery performed [Count of Participants; unit: Participants]
  Vaginal hysterectomy | 21 | 18 | 39
  Salpingectomy | 16 | 14 | 30
  Uterosacral ligament suspension | 16 | 17 | 33
  Sacrospinous ligament suspension | 11 | 13 | 24
  A/P repair | 23 | 20 | 43
  Trachelectomy | 0 | 1 | 1
  Colpocleisis | 3 | 2 | 5
  Vaginal mesh removal | 1 | 0 | 1
  Midurethral sling | 15 | 13 | 28
  Vaginal cuff repair | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scores at 7am After Surgery
Description: Visual analog score: 0 (No pain) - 100 (The worst imaginable pain)
Time Frame: Postoperative day 1 at 7am
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 34 | 31
score on a scale | 29.2 (21.5) | 42.6 (25.8)

2. Secondary Outcome: Visual Analog Scores at Discharge From Post-anesthesia Care Unit
Description: Visual analog score: 0 (No pain) - 100 (The worst imaginable pain)
Time Frame: At the time of discharge from post-anesthesia care unit, on average 1-3 hours from end of surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 34 | 34
score on a scale | 53.1 (26.2) | 56.4 (27.6)

3. Secondary Outcome: Pain Scores 96 Hours After Surgery
Description: Numeric rating pain scale: 0 (No pain) - 100 (The worst imaginable pain)
Time Frame: 96 hours postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 33 | 32
score on a scale | 26.7 (21.8) | 35.5 (24.3)

4. Secondary Outcome: Quality of Recovery Scores on Post op Day 1 (7AM)
Description: Quality of Recovery is a global measure of quality of recovery. It is scored from 40-200. A higher score = better recovery.
Time Frame: 7am on postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 34 | 32
score on a scale | 177.7 (13.95) | 172.3 (18.36)

5. Secondary Outcome: Satisfaction Scores in the Morning After Surgery (7AM)
Description: Satisfaction with overall pain control: 0 (Not satisfied at all) - 100 (Extremely satisfied)
Time Frame: 7am on postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 33 | 31
score on a scale | 81.5 (20.7) | 79.6 (26.8)

6. Secondary Outcome: Satisfaction Scores 96 Hours After Surgery
Description: Satisfaction with overall pain control: 0 (Not satisfied at all) - 100 (Extremely satisfied)
Time Frame: 96 hours postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 33 | 32
score on a scale | 80.5 (26.3) | 79.4 (25.9)

7. Secondary Outcome: Opioid Analgesic Use in the Post-anesthesia Care Unit
Description: Total dose of opioids administered in the post-anesthesia care unit, in morphine equivalents.
Time Frame: Through the time of discharge from the post-anesthesia care unit, on average 1-3 hours from the end of surgery.
Measure: Median (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 36 | 35
morphine milligram equivalents | 5 (7.3) | 7.8 (7.3)

8. Secondary Outcome: Total Postoperative Opioid Use
Description: Total dose of opioids administered (in morphine equivalents) from time of arrival to the post-anesthesia care unit until either they were discharged from the hospital on POD#1 up to 24 hours postop OR if they were discharged on POD#0, the end timepoint was the time of the phone call on POD#1, up to 24 hours after surgery.
Time Frame: From the time a patient arrived in the post-anesthesia recovery unit until discharged from the hospital up to 24 hours OR time of their POD#1 phone call if discharged on same day as surgery up to 24 hours
Measure: Median (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 35 | 34
morphine milligram equivalents | 15 (28.6) | 20.5 (23.9)

9. Secondary Outcome: Severity of Postoperative Non-pain Symptoms
Description: Quality of Recovery Score, Part B "Comfort". Scale 8-40, higher score = better recovery
Time Frame: Postoperative day 1 (7AM)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 34 | 32
score on a scale | 37.2 (3.3) | 35.3 (5.6)

10. Secondary Outcome: Number of Participants With Postoperative Urinary Retention
Description: Incidence of urinary retention
Time Frame: Up to 96 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pudendal Block | Placebo Injection
Number analyzed (Participants) | 36 | 34
Participants | 7 | 4

ADVERSE EVENTS:
Time Frame: Through postop day 4
Arm/Group | Pudendal Block | Placebo Injection
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04198714/Prot_SAP_000.pdf